CLINICAL TRIAL: NCT00001661
Title: Mechanisms of Plasticity in the Human Motor System
Brief Title: Mechanisms of Human Plasticity in the Human System
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970048; 97-N-0048
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-03

CONDITIONS: Blindness; Cerebrovascular Accident; Spinal Cord Injury
Keywords: Plasticity; Use; Stroke; Spinal Cord Injury; Amputation; Intracortical Inhibition
MeSH Terms: conditions — Blindness; Stroke; Spinal Cord Injuries

SUMMARY:
The purpose of this study is to investigate the physiology associated with plasticity of the motor system. Plasticity refers to the process by which neighboring brain cells assume the responsibilities of damaged or diseased brain cells.

The mechanisms behind this process are unknown. However, researchers have several theories about how plastic changes take place. Possible explanations include the growth of new connections between brain cells and the use of previously unused connections.

Researchers plan to use transcranial magnetic stimulation and drug intervention in order to determine the mechanisms responsible for specific types of plasticity.

Previous studies have shown that certain drugs can affect the mechanisms involved in these changes. By using one drug at a time, researchers plan to evaluate the role of each of several different mechanisms in brain reorganization.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the physiology associated with plasticity of the motor system seen in a number of different circumstances. Techniques used will involve the combination of transcranial magnetic stimulation (TMS) and pharmacologic interventions. We propose to use drugs judged to be safe, that either potentiate GABA related intracortical inhibition, change presynaptic release of excitatory aminoacids like glutamate, or decrease the activity of the NMDA receptors (mostly antiepileptic drugs). If plastic changes expressed as larger motor maps or motor evoked potentials (MEP) to TMS are secondary to intracortical disinhibition, administration of a drug that potentiates intracortical inhibition may result in decreased plasticity and smaller motor maps or MEP. This finding would then identify intracortical disinhibition as the mechanism responsible for this type of plasticity. Similarly, if plastic changes decrease with a drug that inhibits release of excitatory aminoacids, or that antagonize the action of NMDA receptors, the mechanism underlying plasticity is likely to be mediated by modulation in the release of excitatory aminoacids or activity in NMDA-receptors.

Results from this study will then provide information about the relative involvement of intracortical disinhibition, modulation in the release of excitatory aminoacids, and role of NMDA receptors in different settings of human plasticity.

ELIGIBILITY:
Must be over 18 years of age.

Must not have personal history of seizures, loss of consciousness, hypertension, psychosis, heart conditions or allergies to any of the drugs.

Women must not be nursing or pregnant.

Patients may have amputations, spinal cord injuries, blindness or large hemispheric lesions from stroke.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260
Dates: Start 1996-12; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cohen LG, Bandinelli S, Findley TW, Hallett M. Motor reorganization after upper limb amputation in man. A study with focal magnetic stimulation. Brain. 1991 Feb;114 ( Pt 1B):615-27. doi: 10.1093/brain/114.1.615. PMID 2004259
- [Background] Ziemann U, Lonnecker S, Steinhoff BJ, Paulus W. Effects of antiepileptic drugs on motor cortex excitability in humans: a transcranial magnetic stimulation study. Ann Neurol. 1996 Sep;40(3):367-78. doi: 10.1002/ana.410400306. PMID 8797526
- [Background] Brasil-Neto JP, Valls-Sole J, Pascual-Leone A, Cammarota A, Amassian VE, Cracco R, Maccabee P, Cracco J, Hallett M, Cohen LG. Rapid modulation of human cortical motor outputs following ischaemic nerve block. Brain. 1993 Jun;116 ( Pt 3):511-25. doi: 10.1093/brain/116.3.511. PMID 8513390